CLINICAL TRIAL: NCT05733637
Title: Validation of a Novel Anxiety Scale (HRAD) During Vascular Access Procedures
Brief Title: HRAD-Vascular Access
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Other Study IDs: 68986
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Anxiety; Vascular Access
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vascular Access: Patients undergo vascular access procedure.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There will be no intervention apply to study participants.

SUMMARY:
The perioperative setting is a common site of pediatric anxiety and distress. Perioperative anxiety in pediatric patients can result in uncooperative behavior, poor postoperative outcomes, and trauma. Given the fast-paced nature of the perioperative environment, many anxiety measures are too time consuming for clinical implementation prior to surgery. Pediatric anesthesiologists need reliable and efficient assessment tools to quickly measure childhood distress to target prophylactic and therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* participants who is undergoing vascular access

Exclusion Criteria:

* Clinically unstable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergo vascular access procedure.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2023-06-11 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Correlation of HRAD± to mYPAS during vascular access procedure | during vascular access procedure
  Correlation between HRAD and mYPAS was assessed by using Fleiss' Kappa. HRAD contains 5-item scale assessing participant's affective state; happy, relaxed, anxious, distressed, with a yes/no answer to cooperation. mYPAS contains 5 items (activity, vocalisation, emotional expressivity, state of apparent arousal, and use of parent). The total score ranges from 0 to 22. Higher scores mean higher levels of anxiety.

SECONDARY OUTCOMES:
Correlation of HRAD± to OBDS-R during vascular access procedure | during vascular access procedure
  Correlation between HRAD and mYPAS was assessed by using Fleiss' Kappa. HRAD contains 5-item scale assessing participant's affective state; happy, relaxed, anxious, distressed, with a yes/no answer to cooperation. OSBD-R contains 8 items (information seeking, crying, screaming, restraint, verbal resistance, emotional support, verbal pain, flail)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Caruso, MD, Study Director — Stanford University
Locations (1):
- Lucile Packard Childrens Hospital Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No